CLINICAL TRIAL: NCT06996067
Title: Essential Coaching Postpartum: Evaluating a Parent-focused Postpartum Text Message Program in Nova Scotia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IWK Health Centre (Other)
Responsible Party: Principal Investigator, Justine Dol, Postdoctoral fellow, IWK Health Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1031429
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Parenting Self-efficacy; Postpartum Anxiety; Postpartum Depression (PPD); Postpartum Stress; Mental Health; Co-parenting Practices
Keywords: text messaging; non-birthing parent; birthing parents; mothers; fathers; digital health
MeSH Terms: conditions — Depression, Postpartum; Psychological Well-Being

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Essential Coaching Postpartum (Experimental)
  Interventions: Behavioral: Essential Coaching Postpartum
- Standard care (No Intervention)

INTERVENTIONS:
Behavioral: Essential Coaching Postpartum — Essential Coaching Postpartum consists of one-way, standardized text messages sent to parents from birth to 6-weeks postpartum to provide evidence-based information on newborn care and mental health. Messages are sent twice a day for the first three weeks (10am and 5pm) and then once a day for the following three weeks (10am), starting the second day after birth.
  Other Names: Essential Coaching for Every Mother; Essential Coaching for Every Partner
  Arms: Essential Coaching Postpartum

SUMMARY:
The transition to parenthood is often an exciting yet hard period for parents. In the first year after a new baby, many parents feel less confident, have more anxiety and depression, and feel more isolated and alone. During this time, many parents use their phones and the Internet to seek out information and support. Thus, we are exploring the opportunity of using mHealth, or mobile health, to provide information directly to parents after the birth of their first baby. We have developed a program for both birthing and non-birthing parents called the Essential Coaching Postpartum program. This program provides 332 parents with text messages sent for 6 weeks after birth to share information on newborn care and parent outcomes. This will be tailored based on whether they are the birthing parent (Essential Coaching for Every Mother) or non-birthing parent (Essential Coaching for Every Partner). We will evaluate this program by comparing a group of parents who receive the messages to a group of parents do not receive any text messages. To determine the success of the Essential Coaching Postpartum program, we will compare parents' confidence, anxiety, depression, and co-parenting between the two groups after six-weeks and six-months. We believe that parents who get the text messages will have higher confidence and co-parenting outcomes and lower anxiety and depression. Our goal with the Essential Coaching Postpartum program is to help make the first few weeks after a new baby less stressful by providing information and support directly to parents that they know they can trust.

ELIGIBILITY:
INCLUSION CRITERIA:

Eligible birthing parents will (1) early postpartum (<7 days) with their first child; (2) understand English; (3) have a cell phone with text and data; and (4) live in Nova Scotia. Eligible non-birthing parents will (1) be early postpartum (<7 days) with their first child; (2) understand English; (3) have a cell phone with text and data; and (4) live in Nova Scotia.

EXCLUSION CRITERIA:

Participants (both birthing and non-birthing parents) will be excluded if: (1) newborn die or are expected to die prior to leaving the hospital; (2) they have no access to mobile phone, either personal or shared; (3) unwilling to receive SMS messages; (4) decline or withdraw to participate; or (5) participated in a previous iteration of this project (e.g., either the development or evaluation).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 332 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Parenting self-efficacy | Enrollment, 6-weeks postpartum, 6-months postpartum
  Parenting self-efficacy will be measured using the Karitane Parenting Confidence Scale (KPCS) tool. This 15-item tool was developed to assess perceived self-efficacy of parents of infants birth to twelve months of age and has acceptable internal consistent (Cronbach's alpha = 0.81) and test-retest reliability (r = 0.88). A cut off score of 39 or less (out of a possible 45) was determine to be a clinically low perceived parenting self-efficacy (PPSE).

SECONDARY OUTCOMES:
Postnatal Anxiety | Enrollment, 6-weeks postpartum, 6-months postpartum
  Postnatal anxiety will be measured using the Postpartum Specific Anxiety Scale (PSAS), a 51-item scale that is a valid and reliable measure to assess anxiety during the first six-months postpartum, with individual factor reliability having a Cronbach's alpha from 0.80 to 0.91 with an overall alpha of 0.95. The optimal cut-off PSAS score for detecting clinical levels of anxiety is 112 with a sensitivity and specificity of 0.75.
Postpartum depression | Enrollment, 6-weeks postpartum, 6-months postpartum
  Postpartum depression will be measured using the 10-item Edinburgh Postnatal Depression Scale (EPDS).. A score above 9 (out of 30) indicating a possibility of postpartum depression 30 in both birthing and non-birthing parents.
Postnatal Childcare Stress | Enrollment, 6-weeks postpartum, 6-months postpartum
  Postpartum stress will be measured using the Postpartum Childcare Stress Checklist, an 18-item scale used to measure parental perceptions of childcare stress in the early postpartum period. Responses are summed to produce a score from 0 to 23, where higher scores indicate a higher level of postpartum childcare stress.
General distress | Enrollment, 6-weeks postpartum, 6-months postpartum
  General distress will be measured using the Depression, Anxiety, and Stress Scale, which is a 21-item scale used to measure the emotional states of depression, anxiety, and stress. High postnatal distress is based on percentile scores, with 0-78 classified as 'normal', 78-87 as 'mild', 87-95 as 'moderate', 95-98 as 'severe', and 98-100 as 'extremely severe'.
Sleep | Enrollment, 6-weeks postpartum, 6-months postpartum
  This will be measured using the PROMIS Short-Form Sleep Related Impairment (4a) and PROMIS Short-Form Sleep Disturbances (4a). Sleep related impairment measures perceptions of alertness, sleepiness, and tiredness during usual waking hours, and the perceived functional impairments during wakefulness associated with sleep problems or impaired alertness. On the other hand, sleep disturbance measures perceptions of sleep quality, sleep depth, and restoration associated with sleep. For the v2.0 adult 4-item form, raw scores range from 4-16, with a corresponding T score. Higher scores indicated higher sleep related impairment and disturbance.
Relationship Satisfaction | Enrollment, 6-weeks postpartum, 6-months postpartum
  This will be measured using the Couple Satisfaction Index-4, which is a 4-item scale used to measure one's satisfaction in a relationship. The CSI-4 contains 4 questions: the first item is scored on a 7-point Likert scale with values from 0 ("Extremely Unhappy") to 6 ("Perfect"), the second is scored on a 6-point Likert scale with values from 0 ("Not at all True") to 5 ("Completely True"), and items 3 and 4 are scored on a 6-point Likert scale with values from 0 ("Not at all") to 5 ("Completely"). A total score is calculated by summing the item responses and ranges from 0 to 21; higher scores are associated with higher levels of satisfaction in the relationship. Scores below 13.5 are associated with notable relationship dissatisfaction.
Co-Parenting | Enrollment, 6-weeks postpartum, 6-months postpartum
  This will be measured using the brief Co-parenting Relationship Scale, which a validated 15-item instrument to assess the five coparenting dimensions of agreement, closeness, child exposure to conflict, coparenting undermining, endorsement of partner's parenting, and labour division.35 Scores range from 0 to 60, with high scores indicating greater coparenting.

CONTACTS AND LOCATIONS:
Locations (1):
- IWK Health, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dol J, Chambers CT, Parker JA, Brooks M, Dennis CL, Seguin D, Goldberg JM, Hughes B, Reese T, Richard G, Calnan K. Effectiveness of the Essential Coaching Postpartum Digital Health Solution on Parenting Self-Efficacy, Mental Health, Well-Being, and Parenting Outcomes: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Oct 17;14:e78209. doi: 10.2196/78209. PMID 41105940